CLINICAL TRIAL: NCT00442221
Title: An Open-Label, Repeat Dose Study Of The Safety Of Combo Formulation In The Treatment Of Multiple Episodes Of Acute Migraine Over 12 Months
Brief Title: The Safety Of Combo Formulation In The Treatment Of Multiple Episodes Of Acute Migraine Over 12 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT400-303
Expanded Access: Available
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Migraine Headaches
Keywords: Migrane headaches
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sumatriptan and Naproxen sodium

SUMMARY:
The objective of this study is to assess the safety of a single-tablet dose of Combo Formulation for the treatment of moderate to severe migraines

DETAILED DESCRIPTION:
The objective of this study is to assess the safety of a single-tablet dose of Combo Formulation for the treatment of moderate to severe migraines, with an optional second dose at least 2 hours following the first dose, if needed. Combo Formulation will be administered on average at least twice per month for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or a female who is not pregnant or is not lactating. A female is eligible to enter and participate in this study if she is of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
   * Child-bearing potential, has a negative pregnancy test (urine or serum) at screen, and employs one of the following acceptable measures of contraception:

     * Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the investigational drug (a minimum of 24 hrs); subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for randomized treatment; or,
     * Female sterilization; or,
     * Sterilization of male partner; or,
     * Implants of levonorgestrel; or,
     * Injectable progestogen; or,
     * Oral contraceptive (combined or progestogen only); or,
     * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or,
     * Any other method with published data showing that the lowest expected failure rate for that method is less than 1% per year.
     * Barrier method only if used in combination with any of the above acceptable methods
2. Subject is 18 - 65 years of age.
3. Subject's first migraine occurred prior to the age of 50 years.
4. Subject has at least a 6-month history, immediately prior to screening, of migraine with or without aura according to the International Headache Society criteria (see Appendix I).
5. Subject experienced an average migraine headache frequency of 2-6 moderate or severe attacks per month in the previous 6 months.
6. Subject is able to distinguish his/her migraine attacks as discrete from any other types of headaches.
7. Subject is willing and able to give written informed consent prior to entry into the study.

Exclusion Criteria:

1. Subject has received another investigational drug within the 4 weeks preceding this study, or subject was enrolled in this study previously.
2. Subject has any concurrent medical or psychiatric condition that may affect the interpretation of efficacy and/or safety data or which otherwise contraindicates participation in a clinical trial with a new chemical entity. This includes, but is not limited to, chronic unstable debilitating diseases such as HIV infection, multiple sclerosis, cancer, etc.
3. Subject has a clinically significant disorder that, in the opinion of the investigator, would result in the subject's inability to understand and comply with the requirements of the study.
4. Subject has a history, symptoms, or signs of ischemic cardiac, cerebrovascular or peripheral vascular syndromes or other significant underlying cardiovascular diseases.
5. Subject has a history of cardiac arrhythmias requiring medication or a history of a clinically significant electrocardiogram (ECG) abnormality that, in the investigator's opinion, contraindicates participation in this study.
6. Subject has a history of cerebrovascular abnormalities including stroke and/or transient ischemic attacks.
7. Subject who, in the investigator's opinion, is likely to have unrecognized cardiovascular disease, based on history or the presence of risk factors (e.g. hypertension, hypercholesterolemia, smoker, obesity, diabetes, strong family history of coronary artery disease, female with surgical or physiological menopause, or male over 40 years of age).
8. Subject has evidence or history of ischemic abdominal syndromes, peripheral vascular disease or Raynaud syndrome.
9. Subject has uncontrolled hypertension at screening (sitting systolic pressure >160 millimeters of mercury (mmHg), diastolic pressure >95 mmHg).
10. Subject has a history of epilepsy or conditions associated with a lowered seizure threshold.
11. Subject has a history of basilar or hemiplegic migraine.
12. Subject has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study; or the subject has any other abnormal laboratory value of clinical significance for this study.
13. Subject has a history of non-migraine (i.e., tension-type, sinus, etc.) headache frequency greater than or equal to 15 days/month in each of the 3 months prior to screening.
14. Subject has had >6 migraine attacks/month in either of the 2 months prior to screening.
15. Subject is currently taking a monoamine oxidase inhibitor (MAOI), has taken a MAOI within the 2 weeks prior to screening, or plans to take a MAOI within 2 weeks after treatment.
16. Subject is currently taking any anti-coagulant (e.g., warfarin) or NSAID (except doses of aspirin ≤325 mg per day being used for cardiovascular prophylaxis) on a regular basis.
17. Subject is currently taking, or has taken in the previous 3 months, a migraine prophylactic medication containing ergotamine, an ergot derivative (dihydroergotamine), or methysergide.
18. Subject is currently taking, or has taken in the previous 4 weeks, herbal preparations containing St. John's Wort (Hypericum perforatum)
19. Subject has hypersensitivity, intolerance, or contraindication to the use of sumatriptan or naproxen sodium, any of its components, or any other 5-HT1 receptor agonist.
20. Subject has a history of allergic reactions to naproxen preparations, including subject in whom aspirin or other NSAID drugs induce the syndrome of asthma, rhinitis, and nasal polyps.
21. Subject is pregnant, actively trying to become pregnant, or breast-feeding.
22. Subject is of childbearing potential and not using adequate contraceptive measures.
23. Subject has a recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence, including the overuse (abuse) of ergotamines and/or narcotics to treat migraines. Ergotamine abuse is daily use for 14 consecutive days or intermittent consumption exceeding 10 mg per week for any two weeks.
24. Subject has participated in an investigational drug trial within the previous four weeks, or plans to participate in another study at any time during the period of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-05; Study Completion 2004-08

PRIMARY OUTCOMES:
END POINTS
Adverse events, physical examination findings, vital signs and clinical laboratory findings will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: David Taylor, Study Director — POZEN
Locations (2):
- United States (2):
  - POZEN Inc., Chapel Hill, North Carolina
  - Headache Wellness Center, Greensboro, North Carolina